CLINICAL TRIAL: NCT01471483
Title: Geriatric Assessment and Nursing Telephone Intervention in Elderly Women With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-164
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Geriatric Assessment; Quality of Life; 11-164; Fallopian Tubes
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patient will receive a phone call from nurse: The proposed study will be a prospective longitudinal feasibility study of 50 older adults with a recent diagnosis of stage II, III or IV ovarian cancer who will receive standard first line chemotherapy and surgery over approximately a six-month period. Half of the 50 patients receive a weekly telephone call from geriatric nurse practitioner (NP); the remaining 25 patients would receive standard oncology care alone (randomization).
  Interventions: Behavioral: geriatric assessment and telephone call from nurse
- patients will not receive a phone call from nurse: The proposed study will be a prospective longitudinal feasibility study of 50 older adults with a recent diagnosis of stage II, III or IV ovarian cancer who will receive standard first line chemotherapy and surgery over approximately a six-month period. Half of the 50 patients receive a weekly telephone call from geriatric nurse practitioner (NP); the remaining 25 patients would receive standard oncology care alone (randomization).
  Interventions: Other: geriatric assessment and no call from nurse

INTERVENTIONS:
Behavioral: geriatric assessment and telephone call from nurse — The geriatric assessment will be completed at four time points: 1) on the day the patient receives a new chemotherapy regimen or within 30 days prior, 2) within 30 days of completion of the chemotherapy regimen (or at 12 months from study entry +/-30 days if the chemotherapy regimen is still being continued), 3) within 30 days prior to surgical debulking, and 4) 30 days after surgical debulking. The patient will receive a phone call once a week by a nurse who is an expert in caring for older patients. He/she will be asking questions about symptoms, medications and support at home. Each call is designed to last less than 30 minutes.
  Groups: patient will receive a phone call from nurse
Other: geriatric assessment and no call from nurse — The geriatric assessment will be completed at four time points: 1) on the day the patient receives a new chemotherapy regimen or within 30 days prior, 2) within 30 days of completion of the chemotherapy regimen (or at 12 months from study entry +/-30 days if the chemotherapy regimen is still being continued), 3) within 30 days prior to surgical debulking, and 4) 30 days after surgical debulking. They will not receive the phone calls, questions and symptoms will be addressed directly by the doctors and nurses on the medical and surgical teams.
  Groups: patients will not receive a phone call from nurse

SUMMARY:
Older woman with ovarian cancer have a worse prognosis compared to younger patients. However, the reason is not known. Currently, the standard of care is to evaluate younger and older patients with cancer the same way. However, older patients with cancer often have more complicated issues to manage. For example, older patients often have other medical problems, take more medications, and be dependent on others for help and transportation. Too often, the medical team is unaware of these issues which can effect the patients care.

The purpose of this study is to apply a set of questions designed specifically for patients with cancer who are older than 65 years of age. These questions are called a geriatric assessment.

The investigators want to better understand which older patients with ovarian cancer will be able to tolerate the chemotherapy and surgery and why. This study will also see if a telephone call from a nurse who specializes in caring for older patients will improve patient care. This study will determine how feasible it is to perform geriatric assessments and telephone calls in patients with ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > or = to age of 65. Will receive platinum-based chemotherapy and surgery at MSKCC for stage II-IV ovarian, fallopian tube or peritoneal cancer.
* Pathologic confirmation or high suspicion based on Ca125 level and/or radiologic evidence of ovarian, fallopian tube or peritoneal cancer.
* Able to understand English.
* Be able to provide informed consent.

Exclusion Criteria:

* Enrolled on a phase I trial.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The MSKCC Gynecologic clinic
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-11-08 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
feasibility of a geriatric assessment (GA) | 2 years
  Geriatric Assessment Measures Selected Based on Reliability, Validity, Brevity, & Prognostic Value. We will measure: the percentage of patients able to complete GA on their own; the length of time to complete GA; patient satisfaction with the GA, identifying items that were distressing or difficult to comprehend; the percentage of patients who completed all four serial GA;
feasibility of a weekly geriatric nursing telephone intervention | 2 years
  the percentage of patients able to complete all weekly telephone calls; the length of time for each telephone call; patient satisfaction with the weekly telephone call.

SECONDARY OUTCOMES:
estimate if the cancer-specific GA parameters will predict toxicity. | 2 years
  describe chemotherapy and surgical toxicity. We will describe the chemotherapy & surgical toxicity, estimate & correlation of toxicity with geriatric assessment variables and determine any differences between the telephone intervention vs. the control groups. We will collect 1) Grade 3-5 chemotherapy toxicity; 2) Hospitalizations; 3) Chemotherapy dose delay or reduction; 4) Percentage of patients who complete all 6 cycles of chemotherapy; 5) Percentage of patients who undergo surgical debulking (optimal, suboptimal, no surgery); 6) Surgical complications (MSKCC GYN Surgical Grading System).
differences in the surgical and chemotherapy toxicity | 2 years
  nursing telephone intervention group vs. the control groups. Will describe chemotherapy & surgical toxicity, estimate any correlation of toxicity with geriatric assessment variables & determine any differences between telephone intervention vs. the control groups. Will collect 1) Grade 3-5 chemotherapy toxicity; 2) hospitalizations; 3) Chemotherapy dose delay or reduction; 4) Percentage of patients who complete all 6 cycles of chemotherapy; 5) Percentage of patients who undergo surgical debulking (optimal, suboptimal, no surgery); 6) Surgical complications (MSKCC GYN Surgical Grading System).

CONTACTS AND LOCATIONS:
Overall Officials: William Tew, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm